CLINICAL TRIAL: NCT04951453
Title: Systemic Nitrosative/Oxidative Stress in Patients with Acute Brain Injury
Acronym: NOX
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of South Wales (Other)
Responsible Party: Principal Investigator, Anton Lund, MD, Rigshospitalet, Denmark
Other Study IDs: H-21004729
Record Dates: First submitted 2021-06-28; First posted 2021-07-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Intracerebral Hemorrhage; Traumatic Brain Injury
Keywords: Nitrosative Stress; Oxidative Stress; Nitric Oxide; Acute Brain Injury; Subarachnoid Hemorrhage; Intracerebral Hemorrhage; Traumatic Brain Injury; Secondary Brain Injury; Neuromonitoring
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebral Hemorrhage; Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (whole blood, serum, plasma, and red blood cells)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Aneurysmal subarachnoid haemorrhage: Patients with SAH (see eligibility criteria below). Planned enrollment: 50 patients.
  Interventions: Other: None (observational)
- Intracerebral haemorrhage: Patients with ICH (see eligibility criteria below). Planned enrollment: 50 patients.
  Interventions: Other: None (observational)
- Traumatic Brain Injury: Patients with TBI (see eligibility criteria below). Planned enrollment: 50 patients.
  Interventions: Other: None (observational)

INTERVENTIONS:
Other: None (observational) — None (observational)

SUMMARY:
Acute brain injury due to traumatic brain injury (TBI), intracerebral haemorrhage (ICH), and aneurysmal subarachnoid haemorrhage (SAH) carries a high morbidity and mortality, in part due to the development of secondary brain injury. The mechanisms behind secondary brain injury are incompletely understood, but oxidative/nitrosative stress and disturbances in the metabolism of the vasodilator nitric oxide (NO) are believed to be involved. The aim of the present study is to characterise systemic changes in markers of oxidative/nitrosative stress and NO metabolism in the early phase after acute brain injury, and to examine their relationship to clinical course, neurological outcome, and mortality.

DETAILED DESCRIPTION:
BACKGROUND:

Acute brain injury due to traumatic brain injury (TBI), intracerebral haemorrhage (ICH), and aneurysmal subarachnoid haemorrhage (SAH) is a major cause of mortality and permanent disability worldwide. Irrespective of its aetiology, acute brain injury is associated with a widespread activation of cellular and biochemical processes which can aggravate the damage after the primary injury - this is termed secondary brain injury.

Nitric oxide (NO) is a potent endogenous vasodilator produced from arginine by the enzyme nitric oxide synthase (NOS), which exists in three isoforms: endothelial, neuronal, and inducible NOS (eNOS, nNOS and iNOS). In conditions of inflammation and oxidative stress (e.g. in acute brain injury), free radicals may react with NO to form peroxynitrite (ONOO-), which is highly reactive and can directly damage biological macromolecules such as lipids and proteins. This phenomenon, i.e. an increased production of reactive nitrogen species potentially leading to cellular damage, is termed nitrosative stress.

It is widely believed that oxidative/nitrosative stress and associated disturbances in the metabolism of NO are involved in the development of secondary brain injury, but the exact role of these mechanisms remains incompletely understood. While some authors believe that NOS dysfunction and a resultant low NO bioavailability is an important cause of secondary brain injury, others argue that an overproduction of NO mediated by iNOS is maladaptive response leading to aggravated tissue injury due to nitrosative stress.

The investigators hypothesise that acute brain injury is associated with an immediate elevation in circulating biomarkers of oxidative stress and a reduction in the bioavailability of NO due to formation of peroxynitrite (nitrosative stress), and that this represents an important mechanism behind the development of secondary brain injury. This decrease in NO availability could contribute to a vicious cycle in which a resulting increase in microvascular resistance, cerebral hypoperfusion, and brain tissue hypoxia further increases free radical production. However, it is further hypothesised that the initial decrease in NO availability is followed by an iNOS-mediated increase in NO metabolites in the subsequent days after injury. The present explorative study will attempt to characterise these changes and their role in patients with acute brain injury.

HYPOTHESES:

1. Patients will have the highest levels of oxidative/nitrosative stress markers and lowest levels of NO metabolites immediately after ictus, with a progressive reduction in oxidative/nitrosative stress markers and increase in NO metabolites over the subsequent days.
2. The degree of oxidative/nitrosative stress will be associated with an unfavourable clinical course (e.g., episodes of neuroworsening), poor neurological outcome, and death.
3. Patients with a higher disease severity (e.g., a higher World Federation of Neurological Surgeons Score for patients with SAH) will have a greater degree of oxidative/nitrosative stress compared to patients with a lower disease severity.
4. The degree of oxidative/nitrosative stress will be associated with the degree of biomarker-determined neurovascular unit injury.
5. The degree of oxidative/nitrosative stress will be associated with evidence of systemic organ dysfunction.
6. The degree of oxidative/nitrosative stress and relative NO-depletion is associated with brain tissue hypoxia, brain metabolic crisis, and cortical spreading depolarisations (in a subset of patients undergoing multimodal neuromonitoring).

METHODS:

The study is a single-center, prospective, explorative, observational study, which will include 50 patients with SAH, 50 patients with ICH, and 50 patients with TBI admitted to the Neurointensive Care Unit (NICU) at Rigshospitalet, Copenhagen. Patient inclusion will continue until the planned number of patients have been enrolled, or until the 1st of May 2023, at which point inclusion will be halted and data will be analysed irrespective of the number of included patients.

Arterial blood samples will be collected at 3 time points: day 0-2 (early), day 3-5 (intermediate) and day 6-8 (late) after admission. If no arterial catheter is available, central venous or peripheral venous samples may be drawn as an alternative. Blood samples will only be collected during admission to the NICU and/or intermediate care unit, and sample collection will be halted in case of discharge to another department.

Demographical, clinical and paraclinical data will be obtained from each patients' electronic medical records. Data from multimodal neuromonitoring (i.e., intracranial pressure, brain tissue oxygenation, cerebral microdialysis, and/or electrocorticography) will be collected continuously along with physiological parameters when available. Neurological outcome (as determined by the modified Rankin Scale) will be determined at 6 months in connection with an outpatient follow-up visit at the hospital or through telephone interviews.

BIOCHEMICAL ANALYSES:

Blood samples will be analysed for the following markers of oxidative stress: the ascorbate radical, lipid hydroperoxides, myeloperoxidase, and the antioxidants glutathione, α/γ-tocopherol, α/β-carotene, retinol and lycopene.

The following NO metabolites will be determined: total plasma NO concentration (nitrate (NO3-) + nitrite (NO2-) + S-nitrosothiols (RSNO)) and total red blood cell bound NO (nitrite (NO2-) + nitrosyl haemoglobin (HbNO) + S-nitrosohaemoglobin (HbSNO)). In addition, 3-nitrotyrosine will be determined as a surrogate marker for peroxynitrite.

The following biomarkers of neurovascular unit injury will be determined: S100ß, glial fibrillary acidic protein, neuron-specific enolase, ubiquitin carboxy-terminal hydrolase L1, neurofilament light-chain and total tau.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Neurointensive Care Unit (NICU) at Rigshospitalet
* Diagnosis of TBI, spontaneous ICH or aneurysmal SAH
* Initiation of blood sampling possible within 3 days after ictus
* Expected length of stay in the NICU and/or intermediate care unit of ≥48 hours
* Closest relatives understand written and spoken Danish

Exclusion Criteria:

* Brain death before inclusion
* Expected death within 24 hours
* ICH secondary to other causes (e.g., a tumour or arteriovenous malformation)
* SAH secondary to other causes (e.g., a mycotic aneurysm or arteriovenous malformation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute brain injury (SAH, ICH or TBI) admitted to the NICU at Rigshospitalet - see detailed inclusion and exclusion criteria above.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome (modified Rankin scale) | 6 months
  Neurological outcome as assessed using the modified Rankin Scale, which measures the degree of disability on a scale from 0 to 6 (higher score indicates a worse outcome)

SECONDARY OUTCOMES:
Mortality | 6 months
  Mortality at 6 months
Neuroworsening | Within 14 days
  Neuroworsening as defined by Morris et al. [1]
Delayed Cerebral Ischaemia (DCI) | Within 14 days
  DCI as defined by Vergouwen et al. [2] (in patients with SAH)

OTHER OUTCOMES:
Levels of brain injury biomarkers | Within 14 days
  Concentrations of the brain injury biomarkers S100ß (μg/L), glial fibrillary acidic protein (pg/mL), neuron-specific enolase (μg/L), ubiquitin carboxy-terminal hydrolase L1 (pg/mL), neurofilament light-chain (pg/mL) and total tau (pg/mL).
Angiographic vasospasm | Within 14 days
  Angiographic vasospasm (in patients with SAH)
Length of stay | During hospitalisation
  Length of stay in the intensive care unit (ICU) and in hospital
Systemic organ dysfunction | During ICU stay
  Systemic organ dysfunction as assessed by the Sequential Organ Failure Assessment (SOFA)-score during stay in the ICU
Brain tissue hypoxia | During ICU stay
  Brain tissue hypoxia (defined as a brain tissue oxygen tension of <20 mmHg) as assessed by invasive brain tissue oxygen monitoring (Integra Licox®) in patients undergoing multimodal neuromonitoring
Brain metabolic crisis | During ICU stay
  Brain metabolic crisis (defined as a lactate/pyruvate ratio >40 with a brain glucose concentration ≤0.7 mmol/L) as assessed by cerebral microdialysis in patients undergoing multimodal neuromonitoring
Cortical spreading depolarisations | During ICU stay
  The frequency (occurrence) of cortical spreading depolarisations as assessed by electrocorticography in patients undergoing multimodal neuromonitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Lund, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data from each individual participant will be available after publication of planned manuscripts, with a valid reason, and after signing a data processing agreement.
Supporting Information: Study Protocol
Time Frame: The approved study protocol will be available upon request until publication of the study results.
Access Criteria: Valid reason and contact with author.

REFERENCES:
- [Background] Morris GF, Juul N, Marshall SB, Benedict B, Marshall LF. Neurological deterioration as a potential alternative endpoint in human clinical trials of experimental pharmacological agents for treatment of severe traumatic brain injuries. Executive Committee of the International Selfotel Trial. Neurosurgery. 1998 Dec;43(6):1369-72; discussion 1372-4. PMID 9848851
- [Background] Vergouwen MD, Vermeulen M, van Gijn J, Rinkel GJ, Wijdicks EF, Muizelaar JP, Mendelow AD, Juvela S, Yonas H, Terbrugge KG, Macdonald RL, Diringer MN, Broderick JP, Dreier JP, Roos YB. Definition of delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage as an outcome event in clinical trials and observational studies: proposal of a multidisciplinary research group. Stroke. 2010 Oct;41(10):2391-5. doi: 10.1161/STROKEAHA.110.589275. Epub 2010 Aug 26. PMID 20798370
- [Background] Stocchetti N, Taccone FS, Citerio G, Pepe PE, Le Roux PD, Oddo M, Polderman KH, Stevens RD, Barsan W, Maas AI, Meyfroidt G, Bell MJ, Silbergleit R, Vespa PM, Faden AI, Helbok R, Tisherman S, Zanier ER, Valenzuela T, Wendon J, Menon DK, Vincent JL. Neuroprotection in acute brain injury: an up-to-date review. Crit Care. 2015 Apr 21;19(1):186. doi: 10.1186/s13054-015-0887-8. PMID 25896893
- [Background] Werner C, Engelhard K. Pathophysiology of traumatic brain injury. Br J Anaesth. 2007 Jul;99(1):4-9. doi: 10.1093/bja/aem131. PMID 17573392
- [Background] Pacher P, Beckman JS, Liaudet L. Nitric oxide and peroxynitrite in health and disease. Physiol Rev. 2007 Jan;87(1):315-424. doi: 10.1152/physrev.00029.2006. PMID 17237348
- [Background] Garry PS, Ezra M, Rowland MJ, Westbrook J, Pattinson KT. The role of the nitric oxide pathway in brain injury and its treatment--from bench to bedside. Exp Neurol. 2015 Jan;263:235-43. doi: 10.1016/j.expneurol.2014.10.017. Epub 2014 Oct 29. PMID 25447937
- [Background] Toda N, Ayajiki K, Okamura T. Cerebral blood flow regulation by nitric oxide: recent advances. Pharmacol Rev. 2009 Mar;61(1):62-97. doi: 10.1124/pr.108.000547. Epub 2009 Mar 16. PMID 19293146
- [Background] Cherian L, Goodman JC, Robertson CS. Brain nitric oxide changes after controlled cortical impact injury in rats. J Neurophysiol. 2000 Apr;83(4):2171-8. doi: 10.1152/jn.2000.83.4.2171. PMID 10758126
- [Background] Sehba FA, Schwartz AY, Chereshnev I, Bederson JB. Acute decrease in cerebral nitric oxide levels after subarachnoid hemorrhage. J Cereb Blood Flow Metab. 2000 Mar;20(3):604-11. doi: 10.1097/00004647-200003000-00018. PMID 10724124
- [Background] Sehba FA, Bederson JB. Nitric oxide in early brain injury after subarachnoid hemorrhage. Acta Neurochir Suppl. 2011;110(Pt 1):99-103. doi: 10.1007/978-3-7091-0353-1_18. PMID 21116923
- [Background] Sobey CG, Faraci FM. Subarachnoid haemorrhage: what happens to the cerebral arteries? Clin Exp Pharmacol Physiol. 1998 Nov;25(11):867-76. doi: 10.1111/j.1440-1681.1998.tb02337.x. PMID 9807657
- [Background] Sehba FA, Chereshnev I, Maayani S, Friedrich V Jr, Bederson JB. Nitric oxide synthase in acute alteration of nitric oxide levels after subarachnoid hemorrhage. Neurosurgery. 2004 Sep;55(3):671-7; discussion 677-8. doi: 10.1227/01.neu.0000134557.82423.b2. PMID 15335435
- [Background] Hino A, Tokuyama Y, Weir B, Takeda J, Yano H, Bell GI, Macdonald RL. Changes in endothelial nitric oxide synthase mRNA during vasospasm after subarachnoid hemorrhage in monkeys. Neurosurgery. 1996 Sep;39(3):562-7; discussion 567-8. doi: 10.1097/00006123-199609000-00026. PMID 8875487
- [Background] Jung CS, Oldfield EH, Harvey-White J, Espey MG, Zimmermann M, Seifert V, Pluta RM. Association of an endogenous inhibitor of nitric oxide synthase with cerebral vasospasm in patients with aneurysmal subarachnoid hemorrhage. J Neurosurg. 2007 Nov;107(5):945-50. doi: 10.3171/JNS-07/11/0945. PMID 17977265
- [Background] Pluta RM. Dysfunction of nitric oxide synthases as a cause and therapeutic target in delayed cerebral vasospasm after SAH. Acta Neurochir Suppl. 2008;104:139-47. doi: 10.1007/978-3-211-75718-5_28. PMID 18456999
- [Background] Bailey DM, Taudorf S, Berg RM, Lundby C, McEneny J, Young IS, Evans KA, James PE, Shore A, Hullin DA, McCord JM, Pedersen BK, Moller K. Increased cerebral output of free radicals during hypoxia: implications for acute mountain sickness? Am J Physiol Regul Integr Comp Physiol. 2009 Nov;297(5):R1283-92. doi: 10.1152/ajpregu.00366.2009. Epub 2009 Sep 2. PMID 19726713